CLINICAL TRIAL: NCT01595711
Title: Prediction of the Occurrence of Chronic Pain After Thoracotomy by Measuring Preoperative Skin Conductance (Pain Monitor Device)
Brief Title: Prediction of Chronic Pain by the Pain Monitor
Acronym: D3C
Status: Terminated | Type: Observational
Why Stopped: Difficulties of recrutment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/37; 2011-A00750-41 (Other: ANSM)
Record Dates: First submitted 2012-04-17; First posted 2012-05-10 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracotomized patients
  Interventions: Device: Pain Monitor

INTERVENTIONS:
Device: Pain Monitor — Measurement of cutaneous conductance

SUMMARY:
The skin conductance algesimeter (Pain Monitor™, Med-Storm Innovation AS, NO-0264 Oslo, Norway)) reflects the sympathetic nervous system by the measurement of the skin conductance of the palm of the hand. SCA detects nociceptive pain fast and continuously, specific to the individual, with higher sensitivity and specificity than other available objective methods.

The skin conductance response to a calibrated noxious stimulus varies among patients. It defines two types of people depending on its magnitude.

The investigators assume that the importance of skin conductance response to a noxious stimulus predicts the occurrence of chronic pain in patients operated by thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sexes
* planned pulmonary resection for cancer performed by a posterolateral thoracotomy
* thoracic epidural analgesia

Exclusion Criteria:

* pregnancy,
* morbid obesity,
* insulin-dependent diabetes with dysautonomia,
* inability to proceed with anesthesia using the BIS signal,
* known allergy to remifentanil, propofol, atracurium or to levobupivacaine,
* contra-indication to nefopam
* contra-indication to ketoprofen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo a lung surgical procedure (thoracotomized patients)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-03-07 (Actual); Primary Completion 2013-09-07 (Actual); Study Completion 2013-09-07 (Actual)

PRIMARY OUTCOMES:
Prediction of chronic pain | one year after surgery
  Prediction of chronic pain by the measurement of skin conductance

SECONDARY OUTCOMES:
Prediction of the postoperative pain | 5 days postoperatively
  Prediction of the postoperative pain by the measurement of skin conductance. Postoperative pain is assessed (pain score) at least twice each day at rest and during mobilisation.
Prediction of the postoperative antalgic requirement | 5 days postoperatively
  Prediction of the postoperative analgesic requirement by the measurement of skin conductance. The analgesic requirement is evaluated by the amount of epidural analgesics.
Prediction of the postoperative antalgic requirement by the genetic study | One year after surgery
  Prediction of the postoperative antalgic requirement by the genetic study
Effect of remifentanil on skin conductance | One hour after anesthesia
  Skin conductance is measured before and after a calibrated noxious stimulus. This test is performed after the induction of anesthesia (propofol) and a first time before remifentanil administration and a second time after.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - CHU Strasbourg, Strasbourg
  - Hopital Foch, Suresnes, Île-de-France Region

REFERENCES:
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532